CLINICAL TRIAL: NCT04323319
Title: The Comparison of the Effects of ESWT and Instrument Assisted Soft Tissue Mobilization Techniques in the Treatment of Chronic Plantar Fasiitis- Randomized Controlled Trial
Brief Title: Comparions the Effect of Different Treatment Modalities on Chronic Plantar Fasiitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bahçeşehir University (Other)
Responsible Party: Principal Investigator, Pelin Pişirici, PT, PHD (c), Lecturer, Bahçeşehir University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: BAP.2018-03.01
Record Dates: First submitted 2019-06-10; First posted 2020-03-26 (Actual); Last update posted 2020-03-26 (Actual); Status verified 2020-03

CONDITIONS: Plantar Fasciitis, Chronic
Keywords: Plantar Fasciitis; Extracorporeal shock wave therapy; Graston Technique; Instrument assisted soft tissue mobilization; Stretching; Plantar pressure analysis
MeSH Terms: conditions — Fasciitis, Plantar

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: There is blind assessor who has 20 year experienced PhD PT. Participants are also blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- ESWT Group (Experimental): Patients in the ESWT group will be treated with ESWT once a week for 4 weeks. Each patient was treated with epine calcaneus and its surroundings. The treatment dose of 10 Hz, 2.5 bar, 2000 shock wave with BTL L-6000 SWT device will be applied by the same therapist. Patient completed plantar fascia and gastrocnemius streching exercises right after treatment. The patient completed the plantar fascia and gastrocnemius stretching exercises right after treatment and also continue at home for 4 weeks, 2 sets per day. Completed 3 repetation for each exercise and stayed in the same position for 30 seconds.
  Interventions: Device: ESWT, Graston Technique
- Graston Technique® Group (Experimental): The application was carried out by Graston Technique® (GT®) certified, a therapist with orthopedic rehabilitation and soft tissue treatments for over 12 years. GT® instruments were used to diagnose and treat the damaged soft tissue of gastrocnemius and plantar fascia. The application protocol and the instruments used according to the regions were determined with reference to the GT® manual. GT® treatment can be given to the same region twice a week. A minimum of 2 days break was given between the applications. Gastrocnemius and plantar fascia application completed in 5 minutes in one leg. GT2, GT4 and GT6 instruments used for application.The patient completed the plantar fascia and gastrocnemius stretching exercises right after treatment and also continue at home for 4 weeks, 2 sets per day. Completed 3 repetation for each exercise and stayed in the same position for 30 seconds.
  Interventions: Device: ESWT, Graston Technique
- Control Group (Experimental): Stretching group was accepted as the control group. the patient monitored once a week at the hospital and continue home stretching program at home. These patients will be given information about plantar fasciitis as well as other groups. Plantar fascia and gastrosoleus self-stretching exercises will be required to be performed twice a day for thirty seconds and three repetitions for 4 weeks. The patients will be followed with an exercise follow-up form.
  Interventions: Device: ESWT, Graston Technique

INTERVENTIONS:
Device: ESWT, Graston Technique — The treatment period for each group was determined as 4 weeks. Stretching program for each group will be given as home exercise program. Stretching exercises will be completed in 3 sets, 2 sets per day, stretching for 30 seconds.
  Graston Technique Group will take treatment 2 times per week, ESWT group will take treatment 1 time per week.
  Other Names: stretching

SUMMARY:
Plantar fasciitis is a common cause of heel pain affecting about 20% of the general population. The basic treatment of plantar fasciitis is conservative. Approximately 85-90% of plantar fasciitis patients can be successfully treated without surgery. Methods include resting, nonsteroidal anti-inflammatory drugs, stretching, shoe orthotics, corticosteroid injections, physical therapy, night splints, and extracorporeal shock wave therapy (ESWT) and ultrasound therapy. Plantar fasciitis treatment is a chronic treatment that has been clearly described in the literature despite the use of treatment modalities. In the literature, treatment modalities which should be used respectively in the treatment of plantar fasciitis are expressed. Nevertheless, it is a chronic disease caused by skipping the treatment steps for various reasons or applying the treatments in the wrong hierarchy. The aim of this project is to compare the effects of stretching exercises, ESWT and instrument-assisted myofascial relaxation technique (Graston Technique®) in the treatment of chronic plantar fasciitis in terms of pain, disability level, quality of life and static and dynamic plantar pressure analysis.

DETAILED DESCRIPTION:
Traditionally, the fascia tissue was described as a single connective tissue surrounding each muscle, muscle fiber and myofibril. In the International Fascia Research Congress held in Vancover, Canada in 2012, the definition of fascia was redefined, including aponeurosis, ligament, tendon, joint capsule, central nervous system, epinerium, bronchial connective tissue and abdominal mesentery. With the emphasis on the importance of fascia in the literature, soft tissue techniques, including fascia, have gained popularity.

Plantar fasciitis is a common cause of heel pain affecting about 20% of the general population. It is usually caused by biomechanical imbalance resulting from tension occurring along the plantar fascia.Plantar fascia is thought to be effective in the pathogenesis of micro-ruptures and inflammation caused by recurrent tension in the insersio. A variety of predisposing factors have also been proposed, including minor trauma, foot pronation, inappropriate shoes, obesity, and prolonged standing. Diagnosis is usually based on clinical history and local sensitivity. The pain is typically felt in the morning and / or after long sitting, in the origin of the plantar aponeurosis, and a centimeter distal to this area, and typically occurs in the first steps after getting out of bed in the morning, resulting in difficulty in daily activities. Basic treatment of plantar fasciitis is conservative. Approximately 85-90% of plantar fasciitis patients can be successfully treated without surgery. Methods include resting, nonsteroidal anti-inflammatory drugs, stretching, shoe additions, orthoses, corticosteroid injections, physical therapy, night splints, and extracorporeal shock wave therapy (ESWT) and ultrasound therapy. Plantar fasciitis treatment is a chronic treatment that has been clearly described in the literature despite the use of treatment modalities.In 2000, the Food and Drug Administration (FDA) approved the use of Extracorporeal Shock Wave Therapy (ESWT), an electrohydraulic device for use in the treatment of chronic plantar fasciitis. Pain, redness, edema and ecchymosis are rarely reported during ESWT treatment, but these effects are not permanent.The exact mechanism of action of the ESWT has not been clearly established. However it is believed that the body responds by increasing the healing ability in that area, by stimulating a repair process. For the patients who treated with ESWT, there was a decrease in pain and an increase in walking ability compared to a control group. ESWT is recommended in chronic plantar fasciitis patients who do not respond to conservative treatment.

Tight bands in the gastrocnemius muscles, myofascial / intramuscular trigger points, may interfere with the development of plantar heel pain. Intramuscular trigger points are defined as hyperirritable areas that are painful on the compression, contraction, or stretching of the muscles in a skeletal muscle stretched and produce pain that is reflected at a distant point away from the intramuscular trigger point, and may affect their stiffness, myofascial constraints and the extensibility of the muscles or fascia.

Instrument-assisted soft tissue mobilization is a treatment approach developed by James Cyriax. Although there are many different name instruments used for myofascial release, the most popular is Graston Technique® (GT®). GT® is a therapeutic technique based on soft tissue mobilization logic, which is used with specially designed instruments and by applying longitudinal pressure along the muscle fibers. This technique differs from conventional cross friction or transverse friction massage. Longitudinal pressure is applied along the fibers of the muscles associated with specially designed instruments. By changing the tissue properties with the instruments, it enables the patient to realize the changing feeling in the treated areas. Damaged tissues are determined by changing the tissue vibration under the instrument. In addition, the clinician's hands with the depth can be much more than the depth that can be brought down and the clinician's fatigue level is reduced. Treatment typically involves greater application at the points of pain than at other tissues.The clinical use of this technique aims to increase the effectiveness of treatment, especially in patients. It is believed that by creating microtrauma in tissue, it will produce a local inflammatory response that promotes the disintegration of scar tissue, opening of adhesions, new collagen synthesis and connective tissue remodeling. The treatment efficacy of the instruments increases the local inflammation response, especially with microtrauma created in the damaged areas, increases the scar tissue destruction, loosens the adhesions, increases collagen synthesis and stimulates the remodeling of the connective tissue.

In the literature, treatment modalities which should be used respectively in the treatment of plantar fasciitis are expressed. Nevertheless, it is a chronic disease caused by skipping the treatment steps for various reasons or applying the treatments in the wrong hierarchy.

The comparison of stress, GT® and the effectiveness of ESWT applications will contribute both to the deficiency of the literature and to decide on effective treatment.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis with plantar fasciitis, between age o 18-60 and have pain for more than 3 months,
* patients with at least 3 conservative treatments were unsuccessful (include usage of anti-inflammatory drugs, cortisone injection and surgical),
* according to Visual Analogue Scale (VAS), patients with (VAS)≥5

Exclusion Criteria:

* calcaneal fracture and implants,
* tarsal tunnel syndrome,
* infection,
* neurological problems,
* tumor,
* coagulated impairments,
* pregnancy

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 63 (Actual)
Dates: Start 2018-12-27 (Actual); Primary Completion 2020-01-30 (Actual); Study Completion 2020-03-01 (Actual)

PRIMARY OUTCOMES:
First step pain: Visuel Analog Scale (VAS) | Changes in the VAS scores of the three groups before the treatment.
  Visuel Analog Scale by using 10 cm likert scale.
First step pain: Visuel Analog Scale (VAS) | Changes in the VAS scores of the three groups 4 weeks after treatment.
  Visuel Analog Scale by using 10 cm likert scale.
First step pain: Visuel Analog Scale (VAS) | Changes in the VAS scores of the three groups 8 weeks after treatment.
  Visuel Analog Scale by using 10 cm likert scale.

SECONDARY OUTCOMES:
Pressure Pain Threshold | Changes in the pressure pain threshold (mean value of three measurement) of the three groups before and 4 weeks after treatment and at 8 weeks will be compared.
  Pressure algometers measure pressure pain thresholds of muscles.Pressure threshold to investigate the effects of both attempts on pain, by a blind assessor evaluated at three points on the affected leg, gastrocnemii (midpoint of the muscle belly), soleus (midpoint of the muscle at 10 cm above the Achilles tendon) on the muscles and on the posterior face of the calcaneus. FDX Force Ten algometer (FDX-Wagner Instruments) is used for evaluation.
Kinesiophobia | Changes in the Tampa scores of the three groups before and 4 weeks after treatment and at 8 weeks will be compared.
  The Tampa Scale for Kinesiophobia (TSK) is a 17 item questionnaire used to assess the subjective rating of kinesiophobia or fear of movement. The range of scores are from 17 to 68 where the higher scores indicate an increasing degree of kinesiophobia.
Foot Function Index | Changes in the Foot function Index scores of the three groups before and 4 weeks after treatment and at 8 weeks will be compared.
  A Foot Function Index (FFI) measures the impact of foot pathology on function in terms of pain, disability and activity restriction.The FFI consists of 23 self-reported items divided into 3 subcategories on the basis of patient values: pain, disability and activity limitation.
  The pain subcategory consists of 9 items and measures foot pain in different situations, such as walking barefoot versus walking with shoes.
  Recorded on a visual analogue scale (VAS), scores range from 0 to 100 mm, with higher scores indicating worse pain. Both total and subcategory scores are calculated.
SF-12 | Pre-intervention, 5th weeks (post-intervention) and 8th weeks.
  SF-12 is composed of 12 subheadings of SF-36. The SF-12 summary scores (PCS-12 and MCS-12) also range from 0 to 100, with higher scores representing better self-reported health.
Plantar Pressure Analysis | Changes in the VAChanges in the Plantar Pressure Analysis of the three groups before and 4 weeks after treatment and at 8 weeks will be compared.
  The platform systems are made of a series of flat, solid pressure sensing elements arranged in a matrix configuration and embedded in the ground to allow normal walking. Platform systems can be used for both static and dynamic applications. With the analyzer sensor medika fm4040 the load distribution of the soles will be evaluated both statically and dynamically.
Global Rating of Change | Global Rating of Change scores will be evaluated at 4 weeks (at the end of treatment) and at 8 weeks.
  General proportion scales provide a flexible, fast and simple method for self-evaluation of improvement in research and clinical settings. provides a way to obtain information on treatment efficacy quickly, flexibly and efficiently. The instrument has advantages such as clinical significance, appropriate reproducibility and sensitivity to change, and is easy to understand by the patient and the practitioner. Scale 11 has a retestability rate of 90% and a minimal clinical significance of 2. In the investigator's study, it was used to evaluate the rate of satisfaction with treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Pelin Pişirici, PT, PhD, Principal Investigator — Medipol University Institute of Health Sciences; Dilber Karagozoglu Coskunsu, PT, PhD, Study Director — Bahçeşehir University Faculty of Health Sciences; Feryal Subaşı, PT, Prof, Study Chair — Yeditepe University Faculty of Health Sciences; Uğur Şaylı, MD. Prof., Study Chair — Yeditepe University Hospital; Elif Tugce Cil, PT, MSc, Study Chair — Yeditepe University Faculty of Health Sciences
Locations (1):
- Pelin Pişirici, Istanbul, Beşiktaş/İstanbul, Turkey (Türkiye)